CLINICAL TRIAL: NCT05221840
Title: A Phase III, Double-blind, Placebo-controlled, Randomised, Multicentre, International Study of Durvalumab Plus Oleclumab and Durvalumab Plus Monalizumab in Patients With Locally Advanced (Stage III), Unresectable Non-small Cell Lung Cancer (NSCLC) Who Have Not Progressed Following Definitive, Platinum-Based Concurrent Chemoradiation Therapy
Brief Title: A Global Study to Assess the Effects of Durvalumab With Oleclumab or Durvalumab With Monalizumab Following Concurrent Chemoradiation in Patients With Stage III Unresectable Non-Small Cell Lung Cancer
Acronym: PACIFIC-9
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9078C00001; 2023-503999-24-00 (Registry Identifier: Clinical Trial Information System (CTIS)); 2021-004346-37 (EudraCT Number)
Record Dates: First submitted 2022-01-14; First posted 2022-02-03 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Locally Advanced NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; monalizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Durvalumab and Oleclumab (Experimental): Durvalumab on Day 1 of each 28-day cycle + Oleclumab on Days 1 and 15 of cycles 1 and 2, then on Day 1 of each subsequent 28-day cycle for up to 12 months
  Interventions: Drug: Durvalumab; Drug: Oleclumab
- Arm B: Durvalumab and Monalizumab (Experimental): Durvalumab + Monalizumab on Day 1 of each 28-day cycle for up to 12 months. Placebo infusion will be administered on Day 15 of cycles 1 and 2 only
  Interventions: Drug: Durvalumab; Drug: Monalizumab; Other: Placebo
- Arm C: Durvalumab and Placebo (Active Comparator): Durvalumab on Day 1 of each 28-day cycle + Placebo on Days 1 and 15 of cycles 1 and 2, then on Day 1 of each subsequent 28-day cycle for up to 12 months
  Interventions: Drug: Durvalumab; Other: Placebo

INTERVENTIONS:
Drug: Durvalumab — Durvalumab IV (intravenous infusion)
Drug: Oleclumab — Oleclumab IV (intravenous infusion)
  Arms: Arm A: Durvalumab and Oleclumab
Drug: Monalizumab — Monalizumab IV (intravenous infusion)
  Arms: Arm B: Durvalumab and Monalizumab
Other: Placebo — Placebo IV (intravenous infusion)
  Arms: Arm B: Durvalumab and Monalizumab; Arm C: Durvalumab and Placebo

SUMMARY:
This is a Phase III, randomised, double-blind, multicentre, international study assessing the efficacy and safety of durvalumab (MEDI4736) in combination with oleclumab (MEDI9447) or durvalumab (MEDI4736) with monalizumab (IPH2201) in adults with locally advanced (Stage III), unresectable NSCLC, who have not progressed following platinum-based cCRT.

ELIGIBILITY:
INCLUSION CRITERIA:

* Participant must be ≥ 18 years at the time of screening.
* Histologically- or cytologically-documented NSCLC and have been treated with concurrent CRT for locally advanced, unresectable (Stage III) disease
* Provision of a tumour tissue sample obtained prior to CRT
* Documented tumour PD-L1 status by central lab
* Documented EGFR and ALK wild-type status (local or central).
* Patients must not have progressed following definitive, platinum based, concurrent chemoradiotherapy
* Participants must have received at least 2 cycles of platinum-based chemotherapy concurrent with radiation therapy
* Participants must have received a total dose of radiation of 60 Gy ±10% (54 Gy to 66 Gy) as part of the chemoradiation therapy, to be randomised. Radiation therapy should be administered by intensity modulated RT (preferred) or 3D-conforming technique.
* WHO performance status of 0 or 1 at randomization
* Adequate organ and marrow function

EXCLUSION CRITERIA:

* History of another primary malignancy except for malignancy treated with curative intent with no known active disease ≥5 years before the first dose of study intervention and of low potential risk for recurrence, adequately resected non-melanoma skin cancer and curatively treated in situ disease, or adequately treated carcinoma in situ or Ta tumours without evidence of disease.
* Mixed small cell and non-small cell lung cancer histology.
* Participants who receive sequential (not inclusive of induction) chemoradiation therapy for locally advanced (Stage III) unresectable NSCLC.
* Participants with locally advanced (Stage III) unresectable NSCLC who have progressed during platinum-based cCRT.
* Any unresolved toxicity CTCAE >Grade 2 from the prior chemoradiation therapy (excluding alopecia).
* Participants with ≥grade 2 pneumonitis from prior chemoradiation therapy.
* History of idiopathic pulmonary fibrosis, drug-induced pneumonitis, or idiopathic pneumonitis - regardless of time of onset prior to randomisation. Evidence of active non-CRT induced pneumonitis (≥ Grade 2), active pneumonia, active ILD, active or recently treated pleural effusion, or current pulmonary fibrosis - diagnosed in the past 6 months prior to randomization.
* Active or prior documented autoimmune or inflammatory disorders (with exceptions)
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1051 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2030-07-02 (Estimated)

PRIMARY OUTCOMES:
Progression Free Surival (PFS) | Up to 5 years after first patient randomized.
  Progression Free Survival (PFS) as assessed by BICR, per RECIST 1.1.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 9 years after first patient randomized
  Overall survival (OS)
Objective response rate (ORR) | Up to 5 years after first patient randomized
  Objective response rate (ORR) per RECIST 1.1 as assessed by BICR
Overall survival (OS) at 24 months | Up to 9 years after first patient randomized
  Overall survival (OS) at 24 months
Duration of response (DoR) | Up to 5 years after first patient randomized
  Duration of response (DoR) per RECIST 1.1 as assessed by BICR
Progression free survival (PFS) at 6, 12, 18, and 24 months | From date of randomization until 24 months
  Progression free survival (PFS) at 6, 12, 18, and 24 months respectively, per RECIST 1.1 as assessed by BICR
Time from randomization to second progression (PFS2) | Up to 5 years after first patient randomized
  Time from randomization to second progression (PFS2)
Time from randomization to first date of distant metastasis or death (TTDM) | Up to 5 years after first patient randomized
  Time from randomization to first date of distant metastasis or death (TTDM)
Time from randomization to start date of first subsequent therapy (TFST) | Up to 9 years after first patient randomized
  Time from randomization to start date of first subsequent therapy (TFST)
Progression free survival (PFS) as assessed by Investigator | Up to 5 years after first patient randomized
  Progression free survival (PFS) as assessed by Investigator
IHC analysis of PD-L1 TC expression | Up to 5 years after first patient randomized
  IHC analysis of PD-L1 TC expression relative to efficacy outcomes
Concentration of Durvalumab | From date of randomization until 3 months after date of last IP dose
  To assess the Pharmacokinetics of Durvalumab when in combination with Monalizumab or Oleclumab - serum peak and trough concentrations
Anti-drug antibodies (ADAs) | From date of randomization until 3 months after date of last IP dose
  The immunogenicity of durvalumab, oleclumab, and monalizumab as assessed by presence of anti-drug antibodies (ADAs)
Time to deterioration in pulmonary symptoms (TTFCD) | Up to 5 years after last patient randomized
  Time to deterioration in pulmonary symptoms (TTFCD)
Concentration of Oleclumab | From date of randomization until 3 months after last dose of IP
  To assess the Pharmacokinetics of Oleclumab when in combination with Durvulumab - serum peak and trough concentrations
Concentration of Monalizumab | From date of randomization until 3 months after last dose of IP
  To assess the Pharmacokinetics of Monalizumab when in combination with Durvalumab - serum peak and trough concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Barlesi, MD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris
Locations (173):
- United States (31):
  - Research Site, San Diego, California
  - Research Site, New Haven, Connecticut
  - Research Site, Stuart, Florida
  - Research Site, Urbana, Illinois
  - Research Site, New Albany, Indiana
  - Research Site, Lexington, Kentucky
  - Research Site, Louisville, Kentucky
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Grand Rapids, Michigan
  - Research Site, Duluth, Minnesota
  - Research Site, Billings, Montana
  - Research Site, Ridgewood, New Jersey
  - Research Site, Ithaca, New York
  - Research Site, Greensboro, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, York, Pennsylvania
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Houston, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Fredericksburg, Virginia
  - Research Site, Richmond, Virginia
  - Research Site, Richland, Washington
  - Research Site, Spokane, Washington
  - Research Site, Tacoma, Washington
  - Research Site, Milwaukee, Wisconsin
- Australia (9):
  - Research Site, Box Hill
  - Research Site, East Melbourne
  - Research Site, Elizabeth Vale
  - Research Site, Gosford
  - Research Site, Heidelberg
  - Research Site, Kogarah
  - Research Site, South Brisbane
  - Research Site, St Albans
  - Research Site, Westmead
- Brazil (11):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Florianópolis
  - Research Site, Fortaleza
  - Research Site, Jaú
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Recife
  - Research Site, São Paulo
  - Research Site, Uberlândia
  - Research Site, Vitória
- Canada (8):
  - Research Site, Edmonton, Alberta
  - Research Site, Barrie, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Rimouski, Quebec
- China (20):
  - Research Site, Anyang
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Kunming
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Nanning
  - Research Site, Nantong
  - Research Site, Neijiang
  - Research Site, Ningbo
  - Research Site, Shaoguan
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Zhanjiang
  - Research Site, Zhengzhou
  - Research Site, Zhongshan
- Colombia (4):
  - Research Site, Barranquilla
  - Research Site, Bogota D.C.
  - Research Site, Medellín
  - Research Site, Valledupar
- France (12):
  - Research Site, Avignon
  - Research Site, Besançon
  - Research Site, Bordeaux
  - Research Site, Clermont-Ferrand
  - Research Site, Créteil
  - Research Site, Lorient
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (9):
  - Research Site, Erfurt
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Esslingen am Neckar
  - Research Site, Georgsmarienhütte
  - Research Site, Gütersloh
  - Research Site, Hanover
  - Research Site, Oldenburg
  - Research Site, Würzburg
- Italy (8):
  - Research Site, Brescia
  - Research Site, Florence
  - Research Site, Lucca
  - Research Site, Meldola
  - Research Site, Orbassano
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Roma
- Japan (11):
  - Research Site, Himeji-shi
  - Research Site, Hiroshima
  - Research Site, Kashiwa
  - Research Site, Kurume-shi
  - Research Site, Natori-shi
  - Research Site, Niigata
  - Research Site, Osaka
  - Research Site, Sendai
  - Research Site, Tokushima
  - Research Site, Toon-shi
  - Research Site, Wakayama
- Research Site, Lima, Peru
- Poland (7):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Koszalin
  - Research Site, Poznan
  - Research Site, Siedlce
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
- Portugal (3):
  - Research Site, Lisbon
  - Research Site, Loures
  - Research Site, Porto
- South Korea (5):
  - Research Site, Changwon-si
  - Research Site, Cheongju-si
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Suwon
- Spain (5):
  - Research Site, Barcelona
  - Research Site, Granada
  - Research Site, Madrid
  - Research Site, Santiago de Compostela
  - Research Site, Valencia
- Taiwan (5):
  - Research Site, Hsinchu
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan
- Thailand (7):
  - Research Site, Bangkok
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Lampang
  - Research Site, Muang
  - Research Site, Mueang
  - Research Site, Naimuang
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Diyarbakır
  - Research Site, Goztepe Istanbul
  - Research Site, Karşıyaka
- United Kingdom (10):
  - Research Site, Belfast
  - Research Site, Bristol
  - Research Site, Dundee
  - Research Site, Edinburgh
  - Research Site, London
  - Research Site, Middlesbrough
  - Research Site, Poole
  - Research Site, Torquay
  - Research Site, Truro
  - Research Site, Wolverhampton
- Vietnam (3):
  - Research Site, Haiphong
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Barlesi F, Cho BC, Goldberg SB, Yoh K, Zimmer Gelatti AC, Mann H, Gopinathan A, Bielecka ZF, Newton M, Aggarwal C. PACIFIC-9: Phase III trial of durvalumab + oleclumab or monalizumab in unresectable stage III non-small-cell lung cancer. Future Oncol. 2024;20(29):2137-2147. doi: 10.1080/14796694.2024.2354160. Epub 2024 Jul 18. PMID 39023287
- See also: Lung Cancer Study Locator details — https://www.lungcancerstudylocator.com/trial/listing/332562